CLINICAL TRIAL: NCT03078244
Title: Protocol for a Multicentre Survey of Patients With Treatment Resistant Hypertension
Acronym: SPIRIT
Status: Completed | Type: Observational
Sponsor: Emerald Clinical Inc. (Industry)
Collaborators: The George Institute (Other); Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: ACHT41
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Treatment Resistant Hypertension
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: N/A, observational study

SUMMARY:
Project aims to determine the number of individuals with treatment resistant hypertension and to define the characteristics of these patients and estimate disease frequency. The study will be a retrospective review of medical record data based upon de-identified information and will require no patient contact.

ELIGIBILITY:
Inclusion Criteria:

* > = 18 years of age
* No known secondary cause of hypertension
* History of uncontrolled hypertension while using 3 or more anti-hypertensive agents
* Controlled blood pressure using 4 or more different anti-hypertensive agents

Exclusion Criteria:

N/A

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with treatment resistant hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Number of adult subjects with treatment resistant hypertension | one year